CLINICAL TRIAL: NCT05001945
Title: A Randomized, Double-blind, Placebo-controlled, Dose-ranging, Multicenter Phase 2 Study to Evaluate the Safety, Efficacy, and Tolerability of MLS-101 in Subjects With Uncontrolled Hypertension
Brief Title: Trial on the Safety and Efficacy of MLS-101 in Patients With Uncontrolled Hypertension
Acronym: Target-HTN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mineralys Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLS-101-201
Record Dates: First submitted 2021-07-20; First posted 2021-08-12 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Hypertension, Renal
Keywords: Blood pressure; Uncontrolled hypertension; Phase II
MeSH Terms: conditions — Hypertension, Renal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Part I) (Placebo Comparator): Placebo tablet(s) by mouth once or twice daily.
  Interventions: Other: Placebo (Part I)
- Dose 1 (Part I) (Experimental): MLS-101 tablet(s) by mouth once or twice daily.
  Interventions: Drug: MLS-101 (Part I)
- Dose 2 (Part I) (Experimental): MLS-101 tablet(s) by mouth once or twice daily.
  Interventions: Drug: MLS-101 (Part I)
- Dose 3 (Part I) (Experimental): MLS-101 tablet(s) by mouth once or twice daily.
  Interventions: Drug: MLS-101 (Part I)
- Placebo (Part II) (Placebo Comparator): Placebo tablet(s) by mouth once daily.
  Interventions: Other: Placebo (Part II)
- Dose (Part II) (Experimental): MLS-101 tablet(s) by mouth once daily.
  Interventions: Drug: MLS-101 (Part II)

INTERVENTIONS:
Drug: MLS-101 (Part I) — MLS-101 tablet(s) by mouth once or twice daily.
  Arms: Dose 1 (Part I); Dose 2 (Part I); Dose 3 (Part I)
Other: Placebo (Part I) — Placebo tablet(s) by mouth once or twice daily.
  Arms: Placebo (Part I)
Other: Placebo (Part II) — Placebo tablet(s) by mouth once daily.
  Arms: Placebo (Part II)
Drug: MLS-101 (Part II) — MLS-101 tablet(s) by mouth once daily.
  Arms: Dose (Part II)

SUMMARY:
A randomized, double-blind, placebo-controlled, dose-ranging, Phase II study to evaluate the safety, efficacy, and tolerability of MLS-101 in Subjects With Uncontrolled Hypertension

ELIGIBILITY:
Inclusion Criteria:

1. Male and nonpregnant, nonlactating female subjects ≥ 18 years of age.
2. Written informed consent Health Insurance Portability and Accountability Act authorization, and local patient privacy required documentation for this study have been obtained
3. Automated office blood pressure (AOBP) with SBP ≥ 130 mm Hg
4. Background antihypertensive treatment of ≥ 2 drugs
5. Serum cortisol ≥ 18 mcg/dL

Exclusion Criteria:

1. Concomitant use of epithelial sodium channel inhibitors or mineralocorticoid receptor antagonists

3. Subjects with hypokalemia

4. Subjects with hyperkalemia

5. Subjects with serum cortisol < 3 mcg/dL

6. Subjects with serum sodium < 135 mEq/L

7. Subjects with estimated glomerular filtration rate < 60 mL/min/1.73m2

8. Subjects with type 1 or uncontrolled (hemoglobin A1c ≥ 9%) type 2 diabetes mellitus

9. Subjects with body mass index > 40 kg/m2

10. Subjects with unstable angina

11. Subjects with SBP ≥ 175 mm Hg or DBP ≥ 100 mm Hg for Part 1 and SBP ≥ 160 mm Hg or DBP ≥ 100 mm Hg for Part 2 at Pre-Screening, Screening/Start of Placebo Run-in, or Randomization

12. Subjects with a decrease in SBP ≥ 20 mm Hg or DBP ≥ 10 mm Hg from sitting to standing position at screening

13. Subjects who, in the opinion of the investigator, have suspected nonadherence to antihypertensive treatment

14. Subjects who, in the opinion of the investigator, have any major medical illness or symptoms

15. Subjects who, in the opinion of the investigator, have any acute or chronic medical or psychiatric condition

16. Subjects undergoing treatment with any of the following medications:

1. Topical corticoids
2. Sympathomimetic decongestants
3. Theophylline
4. Phosphodiesterase type 5 inhibitors
5. NSAIDs
6. Intramuscular steroids
7. Estrogen
8. Cytochromes
9. Strong CYP3A and CYP3A4 inducers

   17. Subjects with known hypersensitivity to MLS-101 or any of the excipients

   18. Subjects who are night-shift workers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-10-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Site 103, Lincoln, California
  - Site 129, Torrance, California
  - Site 135, Tustin, California
  - Site 131, Clearwater, Florida
  - Site 105, Coral Gables, Florida
  - Site 108, Greenacres City, Florida
  - Site 134, Jupiter, Florida
  - Site 146, Miami, Florida
  - Site 137, Miami, Florida
  - Site 139, Miami, Florida
  - Site 143, Miami, Florida
  - Site 122, Pembroke Pines, Florida
  - Site 102, Tampa, Florida
  - Site 118, Albany, Georgia
  - Site 109, Fayetteville, Georgia
  - Site 125, Lawrenceville, Georgia
  - Site 136, Arlington Heights, Illinois
  - Site 138, Bossier City, Louisiana
  - Site 154, Hammond, Louisiana
  - Site 148, Shreveport, Louisiana
  - Site 114, Slidell, Louisiana
  - Site 116, Jefferson City, Missouri
  - Site 121, St Louis, Missouri
  - Site 123, Las Vegas, Nevada
  - Site 141, Jamaica, New York
  - Site 133, Asheboro, North Carolina
  - Site 113, Charlotte, North Carolina
  - Site 130, Fayetteville, North Carolina
  - Site 140, Greensboro, North Carolina
  - Site 104, Morgantown, North Carolina
  - Site 150, Raleigh, North Carolina
  - Site 153, Cleveland, Ohio
  - Site 115, Rapid City, South Dakota
  - Site 107, Chattanooga, Tennessee
  - Site 120, Kingsport, Tennessee
  - Site 152, Nashville, Tennessee
  - Site 151, Arlington, Texas
  - Site 145, Cypress, Texas
  - Site 132, Dallas, Texas
  - Site 124, McKinney, Texas
  - Site 147, Mesquite, Texas
  - Site 126, Pearland, Texas
  - Site 128, Richland Hills, Texas
  - Site 112, Forest, Virginia

REFERENCES:
- [Derived] Laffin LJ, Rodman D, Luther JM, Vaidya A, Weir MR, Rajicic N, Slingsby BT, Nissen SE; Target-HTN Investigators. Aldosterone Synthase Inhibition With Lorundrostat for Uncontrolled Hypertension: The Target-HTN Randomized Clinical Trial. JAMA. 2023 Sep 26;330(12):1140-1150. doi: 10.1001/jama.2023.16029. PMID 37690061

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After successful screening, subjects with plasma renin activity (PRA) ≤1ng/mL/h began a single-blind (SB) run-in period of BID oral treatment with placebo (PBO) in Part 1, and subjects with PRA >1ng/mL/h began a SB QD oral treatment with PBO in Part 2, while continuing on stable doses of background AHT medications. Subjects returned 2 weeks later on Day 1, and those who continued to meet eligibility requirements were randomized in 1:1 fashion with PBO (Part 1), or 6:1 fashion with PBO (Part 2).
Groups:
- Placebo - Part 1: Participants received matching placebo, taken orally, for 8 weeks in Part 1 of the study
- Lorundrostat 12.5 mg BID - Part 1: Participants received 12.5 mg of lorundrostat twice daily, taken orally, for 8 weeks in Part 1 of the study
- Lorundrostat 25 mg BID - Part 1: Participants received 25 mg of lorundrostat twice daily, taken orally, for 8 weeks in Part 1 of the study
- Lorundrostat 12.5 mg QD - Part 1: Participants received 12.5 mg of lorundrostat once daily, taken orally, for 8 weeks in Part 1 of the study
- Lorundrostat 50 mg QD - Part 1: Participants received 50 mg of lorundrostat once daily, taken orally, for 8 weeks in Part 1 of the study
- Lorundrostat 100 mg QD - Part 1: Participants received 100 mg of lorundrostat once daily, taken orally, for 8 weeks in Part 1 of the study
- Placebo - Part 2: Participants received matching placebo, taken orally, for 8 weeks in Part 2 of the study
- Lorundrostat 100 mg QD - Part 2: Participants received 100 mg of lorundrostat once daily, taken orally, for 8 weeks in Part 2 of the study
Period: Overall Study
Arm/Group | Placebo - Part 1 | Lorundrostat 12.5 mg BID - Part 1 | Lorundrostat 25 mg BID - Part 1 | Lorundrostat 12.5 mg QD - Part 1 | Lorundrostat 50 mg QD - Part 1 | Lorundrostat 100 mg QD - Part 1 | Placebo - Part 2 | Lorundrostat 100 mg QD - Part 2
Started | 30 | 22 (Following the completion of the planned interim analysis, the two lowest doses in Part 1 (i.e., 12.5 mg QD and 12.5 mg BID) were dropped from the study and no further subjects were enrolled in these treatment arms.) | 30 | 23 (Following the completion of the planned interim analysis, the two lowest doses in Part 1 (i.e., 12.5 mg QD and 12.5 mg BID) were dropped from the study and no further subjects were enrolled in these treatment arms.) | 28 | 30 | 6 | 31
Completed | 29 | 18 | 28 | 18 | 26 | 27 | 6 | 30
Not Completed | 1 | 4 | 2 | 5 | 2 | 3 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Not completed — Not specified by Investigator | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consisted of all randomized subjects. This analysis set was used for summaries of subject study disposition, with subjects analyzed according to the randomized study treatment group they were assigned to.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - Part 1 | Lorundrostat 12.5 mg BID - Part 1 | Lorundrostat 25 mg BID - Part 1 | Lorundrostat 12.5 mg QD - Part 1 | Lorundrostat 50 mg QD - Part 1 | Lorundrostat 100 mg QD - Part 1 | Placebo - Part 2 | Lorundrostat 100 mg QD - Part 2 | Total
Number analyzed (Participants) | 30 | 22 | 30 | 23 | 28 | 30 | 6 | 31 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (10.7) | 68.1 (10.1) | 64.8 (9.7) | 65.2 (11.3) | 64.7 (9.5) | 68.7 (8.9) | 62.7 (12.3) | 66.6 (10.6) | 65.7 (10.2)
Age, Customized [Count of Participants; unit: Participants]
  <65 | 17 | 6 | 14 | 10 | 15 | 9 | 4 | 8 | 83
  65-79 | 12 | 13 | 15 | 10 | 13 | 17 | 2 | 22 | 104
  >=80 | 1 | 3 | 1 | 3 | 0 | 4 | 0 | 1 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 19 | 12 | 15 | 18 | 4 | 21 | 120
  Male | 13 | 8 | 11 | 11 | 13 | 12 | 2 | 10 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 17 | 10 | 14 | 16 | 2 | 17 | 95
  Not Hispanic or Latino | 18 | 15 | 13 | 12 | 14 | 13 | 4 | 12 | 101
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 16 | 7 | 7 | 11 | 8 | 15 | 2 | 6 | 72
  White | 13 | 15 | 23 | 11 | 19 | 14 | 4 | 25 | 124
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 30 | 22 | 30 | 23 | 28 | 30 | 6 | 31 | 200
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.9 (4.9) | 32 (5.2) | 30.6 (5.5) | 30.6 (4.9) | 32.0 (5.0) | 30.4 (5.5) | 32.0 (3.9) | 30.5 (4.4) | 31.1 (5.0)
Seated Automated Office-measured Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 142.9 (10.7) | 142.6 (13.3) | 142.8 (13.1) | 142.9 (13.7) | 140.0 (12.1) | 142.2 (13.4) | 135.3 (5.5) | 139.8 (9.1) | 141.6 (12.0)
Seated Automated Office-measured Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 83.8 (9.5) | 81.6 (9.4) | 80.1 (9.3) | 80.3 (12.0) | 84.7 (7.0) | 78.5 (10.0) | 81.5 (7.9) | 78.6 (10.0) | 81.1 (9.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Office-measured Systolic Blood Pressure (SBP) at Study Week 8 Compared to Placebo
Description: The primary outcome was defined as the change in office-measured (mean of last 2 of 5 unattended measurements using an automated oscillometric sphygmomanometer device after approximately 5 minutes of rest in the seated position) SBP from baseline to the end of Study Week 8. The primary efficacy analysis was performed using a mixed model repeated measures (MMRM) approach with defined fixed effects per the statistical analysis plan. A least-square estimate of the mean difference between each dose group and the placebo group is provided for Week 8.
Time Frame: 8 Weeks
Population: The full analysis set included all randomized subjects who received at least 1 dose of randomized study treatment (lorundrostat or placebo). Subjects were analyzed according to the randomized study treatment group.
  Per the study SAP, modelled analysis comparisons for Part 2 were performed for 100 mg QD Part 2 vs 100mg QD Part 1, and not to Placebo - Part 2. Accordingly, while subjects were analyzed, modelled LSmeans for Placebo - Part 2 were not reported.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo - Part 1 | Lorundrostat 12.5 mg BID - Part 1 | Lorundrostat 25 mg BID - Part 1 | Lorundrostat 12.5 mg QD - Part 1 | Lorundrostat 50 mg QD - Part 1 | Lorundrostat 100 mg QD - Part 1 | Placebo - Part 2 | Lorundrostat 100 mg QD - Part 2
Number analyzed (Participants) | 29 | 19 | 28 | 19 | 28 | 25 | 0 | 31
mmHg | -4.10 (2.62) | -11.3 (3.15) | -11.07 (2.65) | -5.63 (3.16) | -13.69 (2.67) | -11.92 (2.77) |  | -11.43 (2.41)

2. Secondary Outcome: Change in 24-hour Ambulatory Blood Pressure Monitoring (ABPM) Mean Systolic Blood Pressure (SBP) and Mean Diastolic Blood Pressure (DBP) From Baseline to End of Treatment (EoT)
Description: The ABPM SBP was measured at baseline and EoT. Change in ABPM-derived mean SBP and DBP from baseline to EoT was analyzed using an ANCOVA with a term for treatment group and a baseline mean 24-hour value as a covariate.
Time Frame: 8 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo - Part 1 | Lorundrostat 12.5 mg BID - Part 1 | Lorundrostat 25 mg BID - Part 1 | Lorundrostat 12.5 mg QD - Part 1 | Lorundrostat 50 mg QD - Part 1 | Lorundrostat 100 mg QD - Part 1 | Placebo - Part 2 | Lorundrostat 100 mg QD - Part 2
Number analyzed (Participants) | 26 | 16 | 26 | 15 | 28 | 24 | 0 | 27
mmHg
  Mean SBP | -1.01 (2.38) | -5.78 (3.03) | -9.05 (2.38) | -2.51 (3.15) | -4.86 (2.34) | -6.34 (2.5) |  | -1.02 (2.64)
  Mean DBP | -0.90 (1.46) | -5.14 (1.85) | -6.03 (1.45) | -2.34 (1.91) | -3.64 (1.40) | -6.14 (1.51) |  | -0.07 (1.69)

3. Secondary Outcome: Week 8 Change From Baseline in Office-measured Diastolic Blood Pressure (DBP)
Description: Change in office-measured (average of last 2 of 5 unattended measurements using an automated oscillometric sphygmomanometer device after approximately 5 minutes of rest in the seated position) DBP from baseline to the end of study at week 8.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo - Part 1 | Lorundrostat 12.5 mg BID - Part 1 | Lorundrostat 25 mg BID - Part 1 | Lorundrostat 12.5 mg QD - Part 1 | Lorundrostat 50 mg QD - Part 1 | Lorundrostat 100 mg QD - Part 1 | Placebo - Part 2 | Lorundrostat 100 mg QD - Part 2
Number analyzed (Participants) | 29 | 19 | 28 | 19 | 28 | 25 | 0 | 30
mmHg | -1.63 (1.66) | -5.47 (2.02) | -4.12 (1.68) | -3.76 (2.02) | -7.09 (1.70) | -5.75 (1.77) |  | -5.55 (1.42)

4. Secondary Outcome: Number of Participants With Blood Pressure ≤ 130/80 mmHg at Week 8
Description: Each participant was assessed as a success if the Week 8 value for SBP was ≤130 mmHg and DBP ≤80 mmHg; subjects not meeting both these thresholds were assessed as a failure. Subjects missing an assessment at Week 8 or who received rescue medications were also considered failures.
Time Frame: 8 Weeks
Population: The full analysis set included all randomized subjects who received at least 1 dose of randomized study treatment (lorundrostat or placebo). Subjects were analyzed according to the randomized study treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo - Part 1 | Lorundrostat 12.5 mg BID - Part 1 | Lorundrostat 25 mg BID - Part 1 | Lorundrostat 12.5 mg QD - Part 1 | Lorundrostat 50 mg QD - Part 1 | Lorundrostat 100 mg QD - Part 1 | Placebo - Part 2 | Lorundrostat 100 mg QD - Part 2
Number analyzed (Participants) | 30 | 22 | 30 | 23 | 28 | 30 | 6 | 31
Participants | 7 | 7 | 13 | 6 | 12 | 9 | 3 | 17

ADVERSE EVENTS:
Time Frame: 12 weeks; two weeks for Run-in Phase treatment-emergent adverse events (TEAEs) reporting and ten weeks for on-treatment (i.e., post-randomization) TEAE reporting.
Description: Run-in TEAEs are those that occurred following initiation of study drug dosing in Run-in until initiation of randomized treatment.
  On-treatment TEAES are those that occurred following randomization (Day 1) until 14 days post last dose of study drug in both Part 1 and Part 2.
  Subjects with one or more AEs within a level of MedDRA are counted only once in that level.
Groups:
- Run-in: Participants received placebo, taken orally, for up to 2 weeks in the Run-in phase of the study
Arm/Group | Placebo - Part 1 | Lorundrostat 12.5 mg BID - Part 1 | Lorundrostat 25 mg BID - Part 1 | Lorundrostat 12.5 mg QD - Part 1 | Lorundrostat 50 mg QD - Part 1 | Lorundrostat 100 mg QD - Part 1 | Placebo - Part 2 | Lorundrostat 100 mg QD - Part 2 | Run-in
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/22 | 0/30 | 0/23 | 0/28 | 0/30 | 0/6 | 0/31 | 0/305
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/22 | 0/30 | 2/23 | 0/28 | 0/30 | 0/6 | 1/31 | 0/305
Other Adverse Events (participants affected / at risk) | 7/30 | 13/22 | 18/30 | 16/23 | 10/28 | 16/30 | 1/6 | 19/31 | 8/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Part 1 (N=30) | Lorundrostat 12.5 mg BID - Part 1 (N=22) | Lorundrostat 25 mg BID - Part 1 (N=30) | Lorundrostat 12.5 mg QD - Part 1 (N=23) | Lorundrostat 50 mg QD - Part 1 (N=28) | Lorundrostat 100 mg QD - Part 1 (N=30) | Placebo - Part 2 (N=6) | Lorundrostat 100 mg QD - Part 2 (N=31) | Run-in (N=305)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Part 1 (N=30) | Lorundrostat 12.5 mg BID - Part 1 (N=22) | Lorundrostat 25 mg BID - Part 1 (N=30) | Lorundrostat 12.5 mg QD - Part 1 (N=23) | Lorundrostat 50 mg QD - Part 1 (N=28) | Lorundrostat 100 mg QD - Part 1 (N=30) | Placebo - Part 2 (N=6) | Lorundrostat 100 mg QD - Part 2 (N=31) | Run-in (N=305)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 3 | 1 | 2 | 1 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cortisol decreased (Investigations) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 3 | 0 | 1 | 0 | 5 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 5 | 9 | 6 | 3 | 8 | 0 | 8 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Peripheral Swelling (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Monocyte count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet Count Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count deceased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood corticotrophin decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Following the completion of the planned interim analysis in January 2022, the two lowest doses in Part 1 (i.e., 12.5 mg QD and 12.5 mg BID) were dropped from the study and no further subjects were enrolled in these treatment arms. Accordingly, overall subject numbers in these arms is less than originally planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT05001945/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT05001945/SAP_001.pdf